CLINICAL TRIAL: NCT03957655
Title: Safety and Efficacy of Stem Cells From Human Exfoliated Deciduous Teeth for Treatment of Decompensated Liver Cirrhosis
Brief Title: Safety and Efficacy of SHED for Decompensated Liver Cirrhosis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other); CAR-T (Shanghai) Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhaoshen Li, Prof., Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHED01
Record Dates: First submitted 2019-05-19; First posted 2019-05-21 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Liver Cirrhosis
Keywords: Liver Cirrhosis; stem cell; therapy
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to the randomization results of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHED group (Experimental): SHED transplantation via peripheral vein: 1x10E6 SHEDs/kg body weight administered via peripheral vein at week 0,4,8,12.
  Interventions: Biological: SHED group
- Control (No Intervention): Standard medication for viral hepatitis and cirrhosis

INTERVENTIONS:
Biological: SHED group — 1x10E6 MSCs/kg body weight will be administered via peripheral vein for 4 times at week 0,4,8,12
  Arms: SHED group

SUMMARY:
This study is an prospective, randomized control study. Patients with decompensated cirrhosis will be randomly assigned to receive 4 times of SHED treatment plus standard medical care(treatment）or standard medical care (control). The primary outcome is MELD-Na score. Secondary outcomes are Child-Pugh, liver function, life quality and survival.

DETAILED DESCRIPTION:
At present, there is still no effective treatment for liver cirrhosis, and the use of stem cells for the treatment of cirrhosis has caused great concern.Stem cells from human exfoliated deciduous teeth (SHED) has been shown to be safe and effective for liver diseases. Randomization controlled studies are needed to confirm the long term effect of SHED treatment for liver cirrhosis. The present study aimed to investigate the safety and efficacy of SHED in hepatitis B related liver cirrhosis patients.

This study is an prospective, randomized control study. Patients with decompensated cirrhosis will be randomly assigned to receive 4 times of SHED treatment plus standard medical care(treatment）or standard medical care (control). SHED infusion (1x10E6 cells/kg body weight) via peripheral vein will be given at week 0,4,8,12.The primary outcome is MELD-Na score. Secondary outcomes are Child-Pugh, liver function, life quality and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years
2. HBV-related liver cirrhosis with presentations of decompensation
3. Antiviral treatment with nucleotide drugs for more than half a year and HBV DNA is less than the minimum detection limit;
4. Child-Pugh score B and MELD-Na score≤25
5. Written consent

Exclusion Criteria:

1. Hepatic encephalopathy, hepatorenal syndrome, acute phase of severe hepatitis
2. Child-Pugh score A or C
3. Hepatocellular carcinoma or other malignancies
4. Cirrhosis or liver failure caused by non-Hepatitis B
5. Pregnancy or breastfeeding
6. Severe bacteria infection,coinfection with HIV or other viral hepatitis.
7. History of severe allergy to biological products or history of immunization within half a year
8. Patients or family members refused to participate in the study
9. Drug abuse or alcohol abuse
10. Other candidates who are judged to be not applicable to this study by doctors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-02 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Model for End-Stage Liver Disease (MELD)-Na score | baseline and 4,8,12,16,24 week
  The MELD-Na score is a reliable measure of mortality risk in patients with end-stage liver disease.
  MELD-Na score=3.8ln[bilirubin (mg/dl)]+11.21ln(INR) +9.6ln[creatinine (mg/dl) +6.4* (cause: cholestasis and alcoholic cirrhosis are 0, others are 1) +1.59* (135-Na)

SECONDARY OUTCOMES:
Child-Pugh score | baseline and 4,8,12,16,24 week
  The Child-Pugh score is a scoring system to measure the severity of chronic liver disease inclusive of cirrhosis. The point scores are added up and classified as: class A: 5-6 points class B: 7-9 points class C: 10-15 points
  The score is composed from several categories:
  total bilirubin, μmol/l (mg/dl)<34: 1 point 34-50: 2 points >50: 3 points
  serum albumin, g/l>35: 1 point 28-35: 2 points <28: 3 points
  INR<1.7: 1 point 1.7-2.3: 2 points >2.3: 3 points
  presence of ascites none: 1 point mild: 2 points moderate to severe: 3 points
  presence of hepatic encephalopathy none: 1 point grades I-II : 2 point grades III-IV: 3 point
Changes of liver function | baseline and 4,8,12,16,24 week
  Changes of liver function index such as ALT, AST, ALB, TBIL, PT
Changes of life quality | baseline and 4,8,12,16,24 week
  Changes of life quality as assessed by SF-36
Survival Rate at half of one year | half of one year
  Survival rate at half of one year

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Dr., Study Chair — Changhai Hospital; Chengzhong Li, Dr., Study Director — Changhai Hospital; Lei Xin, Dr., Principal Investigator — Changhai Hospital; Jianya Xue, Dr., Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang D, Zhang H, Liang J, Wang H, Hua B, Feng X, Gilkeson GS, Farge D, Shi S, Sun L. A Long-Term Follow-Up Study of Allogeneic Mesenchymal Stem/Stromal Cell Transplantation in Patients with Drug-Resistant Systemic Lupus Erythematosus. Stem Cell Reports. 2018 Mar 13;10(3):933-941. doi: 10.1016/j.stemcr.2018.01.029. Epub 2018 Mar 1. PMID 29478901
- [Background] Xuan K, Li B, Guo H, Sun W, Kou X, He X, Zhang Y, Sun J, Liu A, Liao L, Liu S, Liu W, Hu C, Shi S, Jin Y. Deciduous autologous tooth stem cells regenerate dental pulp after implantation into injured teeth. Sci Transl Med. 2018 Aug 22;10(455):eaaf3227. doi: 10.1126/scitranslmed.aaf3227. PMID 30135248
- [Background] Ohkoshi S, Hara H, Hirono H, Watanabe K, Hasegawa K. Regenerative medicine using dental pulp stem cells for liver diseases. World J Gastrointest Pharmacol Ther. 2017 Feb 6;8(1):1-6. doi: 10.4292/wjgpt.v8.i1.1. PMID 28217369